CLINICAL TRIAL: NCT07266246
Title: Research Assistant
Brief Title: Effectiveness of Aluminum Foil vs White Linen Reflectors in Phototherapy for Neonatal Hyperbilirubinemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KUBRAN
Record Dates: First submitted 2025-09-23; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Premature; Phototherapy; Neonatal Intensive Care Unit; Neonatal Hyperbilirubinemia; Nursing
MeSH Terms: conditions — Premature Birth; Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group using a white sheet as reflective material in conjunction with phototherapy (Experimental): The three sides of the incubator will be covered with a cardboard panel, cut to fit the incubator dimensions, lined with white linen cloth on the inner surface (length 88 cm, width 47 cm, height 34 cm).
  Interventions: Other: reflective material
- Group Using Aluminum Foil as Reflective Material in Combination with Phototherapy (Experimental): The incubators will be enclosed by a panel covered with aluminum foil on three sides (long side 88 cm, short side 47 cm, height 34 cm).
  Interventions: Other: reflective material
- Group Receiving Standard Single Phototherapy (No Intervention): Infants will receive treatment in accordance with standard phototherapy practice.

INTERVENTIONS:
Other: reflective material — When receiving phototherapy treatment in groups, reflective materials (aluminum foil-coated sheet or white sheet-covered sheet) were placed in the incubators.
  Arms: Group Using Aluminum Foil as Reflective Material in Combination with Phototherapy; Group using a white sheet as reflective material in conjunction with phototherapy

SUMMARY:
Background: Indirect hyperbilirubinemia (IHB) is a common neonatal condition, affecting over 60% of term and 80% of preterm infants. Phototherapy is the most widely used, safe, and non-invasive treatment; however, scattering of phototherapy light decreases treatment efficacy, prolongs therapy duration, and increases the risk of side effects. Reflective materials have been suggested to enhance phototherapy effectiveness, yet studies comparing different reflector types remain limited.

Aim: This study aims to compare the effects of using reflective materials (white cloth or aluminum foil) during phototherapy on total serum bilirubin levels, phototherapy duration, length of hospital stay, vital signs, side effects, and nurses' satisfaction in neonates with physiological IHB.

Methods: This single-center, single-blind, randomized controlled trial will be conducted at Ankara University Faculty of Medicine, Cebeci Neonatal Intensive Care Unit. A total of 81 neonates with gestational age 35-42 weeks and total serum bilirubin levels of 15-20 mg/dl will be randomly assigned into three groups: (1) phototherapy with white cloth reflectors, (2) phototherapy with aluminum foil reflectors, and (3) standard phototherapy (control). Data will be collected using an Introductory Information Form, Daily Follow-up Chart, Side Effect Observation Form, and Nurse Satisfaction Questionnaire. Statistical analyses will include parametric and non-parametric tests based on distribution assumptions, with significance set at p<0.05.

Expected Results: It is hypothesized that the use of reflective materials will result in faster reduction of total serum bilirubin, shorter phototherapy and hospitalization durations, more stable vital signs, fewer side effects, and higher nurse satisfaction compared with standard phototherapy.

Conclusion: The study will provide evidence on the comparative effectiveness of two low-cost reflector materials in enhancing phototherapy outcomes, potentially offering a practical and efficient strategy for neonatal hyperbilirubinemia management.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with total serum bilirubin levels between 15-20 mg/dL
* Gestational age between 35-42 weeks
* Birth weight between 2500-4000 g
* APGAR score of 7-10 at the 1st and 5th minutes after birth
* Fed with breast milk and/or formula
* Written and verbal informed consent obtained from parents
* Neonates who can be reached on the first day of phototherapy treatment

Exclusion Criteria:

* Neonates with Rh incompatibility
* Neonates with ABO incompatibility
* Neonates with any congenital anomaly
* Neonates with asphyxia
* Neonates receiving intensive (double) phototherapy
* Neonates with glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Neonates with serum bilirubin levels close to the exchange transfusion threshold
* Neonates whose parents do not consent to participation in the study

Ages: 36 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Total Serum Bilirubin Level | At baseline (prior to phototherapy), 4 hours after initiation, and at the final assessment before discontinuation of phototherapy (up to 24 hours)
  The difference in total serum bilirubin concentration measured at baseline (before phototherapy), at the 4th hour, and at the last measurement during phototherapy, expressed in mg/dL.

SECONDARY OUTCOMES:
Nurse Satisfaction | Measured once at completion of phototherapy (up to 24 hours after initiation)
  Nurses' satisfaction with the use of reflective materials, assessed using a structured questionnaire.
Adverse Events | Measured once at completion of phototherapy (up to 24 hours after initiation)
  Incidence of phototherapy-related side effects (e.g., dehydration, hyperthermia, hypothermia, diarrhea, skin rash, bronze baby syndrome).
Duration of Phototherapy | Measured once at completion of phototherapy (up to 24 hours after initiation)
  Total duration of phototherapy received by each infant, recorded in hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.